CLINICAL TRIAL: NCT04047173
Title: Radiofrequency Ablation Versus Stereotactic Body Radiotherapy for Recurrent Small Hepatocellular Carcinoma: a Randomized, Open-label, Controlled Trial
Brief Title: RFA Versus SBRT for Recurrent Small HCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, Clinical Pro., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFA vs. SBRT for recurrent HCC
Record Dates: First submitted 2019-08-04; First posted 2019-08-06 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: recurrent small hepatocellular carcinoma; Radiofrequency Ablation; Stereotactic Body Radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; Radiofrequency Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic Body Radiotherapy (SBRT) (Experimental): GTV is defined as the intrahepatic lesion on images. Internal target volume (ITV) is defined as the combined volume of GTVs on 10 respiratory phases. Planning target volume (PTV) is generated by adding a 5-mm margin to the ITV. OARs include liver, kidney, stomach, small intestine, and spinal cord. Normal liver volume is defined as the entire liver minus GTV. Dose constraints to OARs were as follows: mean dose of normal liver < 10 Gy, V15Gy (percentage of the normal liver volume receiving ≥ 15 Gy) < 35%; kidneys Dmean < 6 Gy; esophagus D0.5cc < 21 Gy; stomach D0.5cc < 21 Gy; small intestine D0.5cc < 21 Gy; colon D0.5cc < 24 Gy; heart D0.5cc < 30 Gy; ribs D0.5cc < 39 Gy; and spinal cord Dmax < 18 Gy. SBRT is planned using volumetric arc therapy techniques with a prescription dose of 36-54 Gy in 3 fractions, irradiated every other day, and completed within one week. Cone-beam CT is performed before each treatment.
  Interventions: Radiation: stereotactic body radiotherapy (SBRT)
- Radiofrequency Ablation (RFA) (Active Comparator): RFA is performed under intravenous, epidural, or general anesthesia guided by computed tomography (CT) or ultrasound, preferably through a percutaneous or laparoscopic approach. The ablation electrode is precisely inserted into the center of the tumor and ablated at 30-50W power for 5-10 minutes depending on the size and shape of the tumor. Adequate coverage of the tumor lesion with a defined "safety margin" is ensured during ablation. After the completion of tumor ablation, the instrument will remaine active as the electrode is retracted, facilitating needle tract ablation. Contrast-enhanced CT, MRI, and ultrasonography will be performed one month after RFA to detect residual disease. Patients with confirmed complete ablation will undergo periodic follow-up, whereas those with residual tumors undergo repeat RFA procedures. Persistent tumor residue after two consecutive RFA sessions is deemed a treatment failure, and RFA treatment will be discontinued.
  Interventions: Procedure: Radiofrequency ablation (RFA)

INTERVENTIONS:
Radiation: stereotactic body radiotherapy (SBRT) — Radiotherapy dose is 36-54 Gy, irradiated in 3 times, every other day, completed within 1 week.
  Arms: Stereotactic Body Radiotherapy (SBRT)
Procedure: Radiofrequency ablation (RFA) — RFA with a safe margin, RFA again if residual, no more than 2 times.
  Arms: Radiofrequency Ablation (RFA)

SUMMARY:
Recurrence rate of hepatocellular carcinoma (HCC)after resection is as high as 65.0%-83.7%.The recurrence of HCC is the most important factor affecting prognosis. Reasonable and effective treatment of recurrent lesion can significantly improve the long-term treatment efficacy of HCC. The recurrent lesion is usually detected when it's small and is the best indication for local treatment. Local ablation therapy represented by radiofrequency ablation (RFA) is one of the main treatments for recurrent small HCC. Our previous study showed that for recurrent small HCC(≤5cm), RFA has the efficacy equivalent to re-excision, with the advantages of small trauma, quick recovery, low cost, and high quality of life. With the advancement of radiotherapy equipment and the development of precise radiotherapy technology, stereotactic radiotherapy (SBRT) has become one of the routine treatments for HCC, especially for small HCC. Retrospective controlled studies have shown that SBRT is similar to RFA in treating small HCC, and the local control rate may be better than RFA. This project is to conduct a prospective, open, randomized, controlled clinical study of RFA versus SBRT for the treatment of recurrent small hepatocellular carcinoma (single lesion ≤ 5 cm, without extra-hepatic metastasis or vascular invasion). The primary endpoint is local progression-free survival (LPFS), and secondary endpoints are progression-free survival (PFS), overall survival (OS), local control rate (LCR), and safety. Data analysis will be performed according to intention-to-treat (ITT) principles. Subgroup analyses will be conducted according to the predefined stratification factor (tumor diameter ≤ 2 cm vs. 2-5 cm) and other baseline characteristics. The results of these study will help to further improve the long-term treatment efficacy of HCC and establish a rational and effective treatment model for HCC.

DETAILED DESCRIPTION:
Recurrence rate of hepatocellular carcinoma (HCC)after resection is as high as 65.0%-83.7%.The recurrence of HCC is the most important factor affecting prognosis. Reasonable and effective treatment of recurrent lesion can significantly improve the long-term treatment efficacy of HCC. Resection is the preferred treatment for recurrent HCC. Although liver surgery has been progressing in recent years, the alteration of anatomical structure after the first operation, the reduction of liver volume, and the mostly multi-centered origin recurrent lesions, lead to low surgical resection rate, difficult operation, high risk, multiple complications, and high recurrence rate of resection surgery. Salvage liver transplantation is difficult to apply widely due to donor shortages and other problems.

Local ablation, represented by radiofrequency ablation (RFA), is the third major treatment for liver cancer after surgical resection and transcatheter arterial chemoembolization (TACE). Many studies， by us and domestic and foreign scholars， have shown that the long-term efficacy of RFA in the treatment of small HCC is close to that of surgical resection, with a 5-year survival rate of 50%-60%. Therefore，RFA has been recommended as a frontline treatment for small HCC by many international guidelines. The recurrent lesion is usually detected when it's small and is the best indication for RFA. Our previous study showed that for recurrent small HCC(≤5cm), RFA has the efficacy equivalent to re-excision, with the advantages of small trauma, quick recovery, low cost, and high quality of life.

With the development of radiotherapy equipment and the precision imaging technology, especially the emergence of stereotactic radiotherapy (SBRT), the status of radiotherapy in the treatment of HCC is increasing. SBRT is defined as the use of external irradiation technology, which is divided into several fractions, and the high dose of radiotherapy is accurately delivered into the tumor. As a result, tumor is subjected to high dose and the normal tissue around the tumor is exposed to relatively low dose. Compared with conventional fractionated radiotherapy (CRT), SBRT possessed fewer segmentation times (1 to 6 F), higher fractional doses (5 to 20 Gy), and steeper gradients at the edge of the target region, so it has stronger biological effect. Meanwhile, SBRT can also protect the normal organs better, especially for the radiotherapy of smaller tumors. Multiple clinical studies and meta-analyses have shown that SBRT is superior to traditional CRT in the treatment of HCC, and the side effects are lower in the acute phase. SBRT has become a mainstream technology for HCC, and has been recommended as a routine local treatment for HCC by National Comprehensive Cancer Network (NCCN) guidelines and NCI radiotherapy guidelines.

Both RFA and SBRT have been recommended by the NCCN guidelines as a routine local treatment for liver cancer. They are also widely used in the treatment of liver cancer, and their therapeutic efficacy and safety have been widely approved. However, which treatment of recurrent small HCC is superior is still unknown.This project is to conduct a prospective, open, randomized, controlled clinical study of RFA versus SBRT for the treatment of recurrent small HCC (single lesion ≤ 5 cm, without extra-hepatic metastasis or vascular invasion). The primary endpoint is local progression-free survival (LPFS), and secondary endpoints are progression-free survival (PFS), overall survival (OS), local control rate (LCR), and safety. Data analysis will be performed according to intention-to-treat (ITT) principles. Subgroup analyses will be conducted according to the predefined stratification factor (tumor diameter ≤ 2 cm vs. 2-5 cm) and other baseline characteristics. The results of these study will help to further improve the long-term treatment efficacy of HCC and establish a rational and effective treatment model for HCC.

Patients enrolled in this clinical trail received either SBRT or RFA depending on the randomization allocation. Eligible subjects are stratified by maximum tumor diameter (≤ 2 cm vs. 2-5 cm) and randomly assigned in a 1:1 ratio to receive either SBRT or RFA using a computer-generated random assignment system.

As for SBRT group, the treatment follows the protocol below.Immobilization: Patients are immobilized with vacuum bags or styrofoam in the supine position, with the arms raised above the head. 4 dimensional computed tomography (4DCT) scanning: Simple breathing training is conducted before simulation, so that the patient can keep breathing quietly and evenly. A plastic box with reflective marker is placed on the patient's anterior abdominal surface where the respiratory amplitude is relatively large, approximately midway between the xiphoid and the umbilicus. The movement of the marker is recorded by an infrared camera, which is converted into breathing curve by computer software. After the breathing curve becomes stable, the CT data of different respiratory phases is collected by 4DCT in axial cine mode. CT scanning region: From 3-4 cm above the diaphragm to the 4th lumbar vertebra. The intravenous contrast is administered during CT scanning and the slice thickness is 3.0 mm. After 4DCT scanning, images are sorted into 10 phases by the software. Each respiratory cycle is divided into 10 respiratory phases. Delineation of the target volumes and organs at risk: Gross tumor volume (GTV) and organs at risk (OARs) are contoured on the 20% CT image (mid-exhalation). Then the GTV is registered to the other respiratory phases of 4DCT scan by a physicist using Atlas-based Auto-segmentation (ABAS, Electa CMS), and the target volumes are modified and confirmed by a radiation oncologist using the standard window/level settings. GTV is defined as the intrahepatic lesion on images. Internal target volume (ITV) is defined as the combined volume of GTVs on 10 respiratory phases. Planning target volume (PTV) is generated by adding a 5-mm margin to the ITV. OARs include liver, kidney, stomach, small intestine, and spinal cord. Normal liver volume is defined as the entire liver minus GTV. Dose constraints to OARs were as follows: mean dose of normal liver < 10 Gy, V15Gy (percentage of the normal liver volume receiving ≥ 15 Gy) < 35%; kidneys Dmean < 6 Gy; esophagus D0.5cc < 21 Gy; stomach D0.5cc < 21 Gy; small intestine D0.5cc < 21 Gy; colon D0.5cc < 24 Gy; heart D0.5cc < 30 Gy; ribs D0.5cc < 39 Gy; and spinal cord Dmax < 18 Gy. SBRT is planned using volumetric arc therapy techniques with a prescription dose of 36-54 Gy in 3 fractions, irradiated every other day, and completed within one week. Cone-beam CT is performed before each treatment.

As for RFA group, RFA is performed under intravenous, epidural, or general anesthesia guided by computed tomography (CT) or ultrasound, preferably through a percutaneous or laparoscopic approach. The ablation electrode is precisely inserted into the center of the tumor and ablated at 30-50W power for 5-10 minutes depending on the size and shape of the tumor. Adequate coverage of the tumor lesion with a defined "safety margin" is ensured during ablation. After the completion of tumor ablation, the instrument will remaine active as the electrode is retracted, facilitating needle tract ablation. Contrast-enhanced CT, MRI, and ultrasonography will be performed one month after RFA to detect residual disease. Patients with confirmed complete ablation will undergo periodic follow-up, whereas those with residual tumors undergo repeat RFA procedures. Persistent tumor residue after two consecutive RFA sessions is deemed a treatment failure, and RFA treatment will be discontinued.

After the local progression of the tumor, surgical treatment or other treatment methods are considered according to the specific condition.

This study is expected to complete enrollment in 2 years and to follow up for 2 years. The primary analysis is performed in the intention-to-treat population. Kaplan-Meier curves will be used to describe the patient's local recurrence-free survival, and the corresponding statistical dates are calculated, such as median local progression-free survival (LPFS) and bilateral 95% confidential interval(CI). The secondary analysis used hypothesis test and two-sided 95% CIs to compare the time of first local recurrence. Kaplan-Meier curves will also be used to describe the patient's disease progression, and calculated the corresponding statistical data, such as the median overall survival(OS) and bilateral 95% CIs. Logistic regression was used to calculate the odds ratios (OR) for LCR. Subgroup analyses were conducted according to the predefined stratification factor (tumor diameter ≤ 2 cm vs. 2-5 cm) and other baseline characteristics. Safety assessments will be also performed by comparing adverse events in the two groups of patients.

ELIGIBILITY:
Inclusion criteria

1. Aged 18-75 years;
2. Diagnosed with HCC: The diagnosis of HCC will be confirmed according to the " Chinese Guidelines for the Diagnosis and Treatment of Hepatocellular Carcinoma (2019 Edition) " formulated by the National Health Commission of China and the Barcelona Clinic Liver Cancer (BCLC) strategy for prognosis prediction and treatment recommendation of the European Association for the Study of the Liver (EASL);
3. Recurrent small HCC: Single hepatocellular carcinoma ≤ 5 cm that recurs after previous curative resection or thermal ablation, with the recurrence time ≥ 3 months from resection/ablation, and without extrahepatic metastasis or vascular invasion at recurrence;
4. No contraindications for RFA and SBRT treatment;
5. Karnofsky performance score (KPS) ≥ 90;
6. Liver function Child-Pugh class A;
7. Normal liver volume greater than 800 cm3;
8. Expected survival time longer than 6 months;
9. The function of important organs meets the following requirements: a. white blood cell ≥ 3×109/L; b. hemoglobin ≥ 80 g/L; c. platelets ≥ 50×109/L; d. blood creatinine ≤ 1.5 times the upper limit; e. prothrombin time (PT) ≤ 3 seconds above control;
10. Subject has signed the informed consent form and agreed to the treatment and follow-up schedules according to this protocol;
11. Subject must have the ability to understand and voluntarily sign the written informed consent form prior to starting any specific procedure in the study.

Exclusion criteria

1. Presence of extrahepatic metastasis or intrahepatic vascular invasion;
2. More than one recurrent lesion, or maximum diameter > 5 cm;
3. Concomitant severe cardiac, pulmonary, renal, or other major organ dysfunction, severe infection or other comorbidities, unable to tolerate treatment;
4. History of other malignancies;
5. History of allergic reactions to relevant drugs;
6. History of organ transplantation;
7. During pregnancy or lactation;
8. Unable to undergo one of the treatments (RFA or SBRT);
9. Concomitantly receiving other anti-tumor therapy (including immunotherapy and targeted therapy);
10. Other factors that may affect patient enrollment and evaluation results;
11. Refusal to comply with the study protocol requirements for follow-up and refusal to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Local progression-free survival (LPFS) | From date of randomization until the date of first documented local tumor progression or date of death from any cause, whichever came first, assessed up to 2 years.
  LPFS is defined as the time from randomization to local tumor progression or death from any cause. Local tumor progression was defined as progressive disease occurring within 1 cm of the margin of the ablation region or within 1 cm of the margin of the PTV for SBRT.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization until the date of first documented tumor progression or date of death from any cause, whichever came first, assessed up to 2 years.
  PFS is defined as the time from randomization to tumor progression or death from any cause. Tumor progression included local progression, intra-hepatic distant progression (intra-hepatic recurrence beyond the RFA/SBRT target area), and extra-hepatic metastasis.
Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 2 years.
  OS is defined as the time from randomization to death from any cause.
1-,2-,and 3-year local control rate (LCR) | 1, 2, or 3 years after treatment completion.
  The 1-, 2-, and 3-year LCR are defined as the proportion of patients without local failure, tumor growth, or regrowth within 1 cm from the margin of the ablation region or 1 cm from the margin of the PTV for SBRT according to the mRECIST criteria after 1, 2, or 3 years of follow-up.
Safety and adverse events | Acute complications are defined as adverse events occurring within 90 days after treatment; late complications are defined as adverse events occurring after 90 days of treatment completion.
  Treatment-related adverse events are evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (CTCAE 4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Yao-Jun, MD., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Background] Feng K, Yan J, Li X, Xia F, Ma K, Wang S, Bie P, Dong J. A randomized controlled trial of radiofrequency ablation and surgical resection in the treatment of small hepatocellular carcinoma. J Hepatol. 2012 Oct;57(4):794-802. doi: 10.1016/j.jhep.2012.05.007. Epub 2012 May 23. PMID 22634125
- [Background] Ng KKC, Chok KSH, Chan ACY, Cheung TT, Wong TCL, Fung JYY, Yuen J, Poon RTP, Fan ST, Lo CM. Randomized clinical trial of hepatic resection versus radiofrequency ablation for early-stage hepatocellular carcinoma. Br J Surg. 2017 Dec;104(13):1775-1784. doi: 10.1002/bjs.10677. Epub 2017 Nov 1. PMID 29091283
- [Background] Lencioni R, Crocetti L. Local-regional treatment of hepatocellular carcinoma. Radiology. 2012 Jan;262(1):43-58. doi: 10.1148/radiol.11110144. PMID 22190656
- [Background] Lau WY, Leung TW, Yu SC, Ho SK. Percutaneous local ablative therapy for hepatocellular carcinoma: a review and look into the future. Ann Surg. 2003 Feb;237(2):171-9. doi: 10.1097/01.SLA.0000048443.71734.BF. PMID 12560774
- [Background] Tateishi R, Shiina S, Teratani T, Obi S, Sato S, Koike Y, Fujishima T, Yoshida H, Kawabe T, Omata M. Percutaneous radiofrequency ablation for hepatocellular carcinoma. An analysis of 1000 cases. Cancer. 2005 Mar 15;103(6):1201-9. doi: 10.1002/cncr.20892. PMID 15690326
- [Background] Chen MS, Li JQ, Zheng Y, Guo RP, Liang HH, Zhang YQ, Lin XJ, Lau WY. A prospective randomized trial comparing percutaneous local ablative therapy and partial hepatectomy for small hepatocellular carcinoma. Ann Surg. 2006 Mar;243(3):321-8. doi: 10.1097/01.sla.0000201480.65519.b8. PMID 16495695
- [Background] Andolino DL, Johnson CS, Maluccio M, Kwo P, Tector AJ, Zook J, Johnstone PA, Cardenes HR. Stereotactic body radiotherapy for primary hepatocellular carcinoma. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e447-53. doi: 10.1016/j.ijrobp.2011.04.011. Epub 2011 Jun 7. PMID 21645977
- [Background] Bujold A, Massey CA, Kim JJ, Brierley J, Cho C, Wong RK, Dinniwell RE, Kassam Z, Ringash J, Cummings B, Sykes J, Sherman M, Knox JJ, Dawson LA. Sequential phase I and II trials of stereotactic body radiotherapy for locally advanced hepatocellular carcinoma. J Clin Oncol. 2013 May 1;31(13):1631-9. doi: 10.1200/JCO.2012.44.1659. Epub 2013 Apr 1. PMID 23547075
- [Background] Yoon SM, Lim YS, Park MJ, Kim SY, Cho B, Shim JH, Kim KM, Lee HC, Chung YH, Lee YS, Lee SG, Lee YS, Park JH, Kim JH. Stereotactic body radiation therapy as an alternative treatment for small hepatocellular carcinoma. PLoS One. 2013 Nov 8;8(11):e79854. doi: 10.1371/journal.pone.0079854. eCollection 2013. PMID 24255719
- [Background] Sanuki N, Takeda A, Oku Y, Mizuno T, Aoki Y, Eriguchi T, Iwabuchi S, Kunieda E. Stereotactic body radiotherapy for small hepatocellular carcinoma: a retrospective outcome analysis in 185 patients. Acta Oncol. 2014 Mar;53(3):399-404. doi: 10.3109/0284186X.2013.820342. Epub 2013 Aug 21. PMID 23962244
- [Background] Kimura T, Aikata H, Takahashi S, Takahashi I, Nishibuchi I, Doi Y, Kenjo M, Murakami Y, Honda Y, Kakizawa H, Awai K, Chayama K, Nagata Y. Stereotactic body radiotherapy for patients with small hepatocellular carcinoma ineligible for resection or ablation therapies. Hepatol Res. 2015 Apr;45(4):378-86. doi: 10.1111/hepr.12359. Epub 2014 Jun 16. PMID 24849379
- [Derived] Xi M, Yang Z, Hu L, Fu Y, Hu D, Zhou Z, Liu M, Zhao J, Shen J, Li Q, Chen B, Xu L, Fang A, Chen M, Liu S, Zhang Y. Radiofrequency Ablation Versus Stereotactic Body Radiotherapy for Recurrent Small Hepatocellular Carcinoma: A Randomized, Open-Label, Controlled Trial. J Clin Oncol. 2025 Mar 20;43(9):1073-1082. doi: 10.1200/JCO-24-01532. Epub 2024 Dec 18. PMID 39693584